CLINICAL TRIAL: NCT04106570
Title: Neuromuscular Plasticity in Response to Obesity: Effects of Mechanical Overload, Metabolic Disorders and Age
Acronym: PLANEUROB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: AME2P Laboratory, Clermont Auvergne University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2019 BOIRIE 3 (Planeurob); 2019-A00788-49 (Other: 2019-A00788-49)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Obese; Torque production; Neuromuscular fatigue; Electrical muscle stimulation; Knee extensors; Metabolic disorders
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- YOMH (Experimental): Young obese metabolically healthy Description: Aged from 20 to 40 years old and with a glycemia < 1g/l and a triglyceridemia < 1,5g/l.
  Interventions: Other: fatiguability of the knee extensors
- YOMD (Experimental): Young obese with metabolic disorders
  Description: Aged from 20 to 40 years old and with a glycemia > 1g/l and a triglyceridemia > 1,5g/l.
  Interventions: Other: fatiguability of the knee extensors
- MAOMH (Experimental): Middle-Age obese metabolically healthy
  Description: Aged from 40 to 50 years old and with a glycemia < 1g/l and a triglyceridemia < 1,5g/l.
  Interventions: Other: fatiguability of the knee extensors
- MAOMD (Experimental): Middle-Age obese with metabolic disorders Description: Aged from 40 to 50 years old and with a glycemia > 1g/l and a triglyceridemia > 1,5g/l.
  Interventions: Other: fatiguability of the knee extensors
- EOMH (Experimental): Elderly obese metabolically healthy
  Description: Aged from 50 to 70 years old and with a glycemia < 1g/l and a triglyceridemia < 1,5g/l.
  Interventions: Other: fatiguability of the knee extensors
- EOMD (Experimental): Elderly obese with metabolic disorders
  Description: Aged from 50 to 70 years old and with a glycemia > 1g/l and a triglyceridemia > 1,5g/l.
  Interventions: Other: fatiguability of the knee extensors

INTERVENTIONS:
Other: fatiguability of the knee extensors — fatiguability of the knee extensors (in N.m) measured with a dynamometer.

SUMMARY:
Obese people suffer from significant functional limitations, which affect their quality of life and limit their physical activity level. Functional abilities are largely determined by neuromuscular properties, i.e the ability to produce a torque or a power, and fatigability, i.e the ability to maintain a high level of torque production during repeated contractions. Our previous studies on "healthy" obese adolescents (i.e without inflammation or metabolic disorder) suggests that obesity has positive effects on the neural and muscular factors responsible for torque production, with chronic overload acting as a strength training . However, this high torque level is associated with higher fatigability. These results are in contrast with the data obtained on adult obese patients (young and elderly), in whom torque production and fatigability appear to be more impaired, probably due to the development of metabolic disorders associated with obesity (inflammation, insulin resistance and lipid infiltration in muscle) and aging. The respective effects of mechanical overload, metabolic disorders (insulin resistance and lipid infiltration) and aging on neural and muscular factors of torque production and neuromuscular fatigue etiology are not currently known in young adult obese of elderly. Their relationship to the clinical symptoms of mobility troubles is also unknown. However, this knowledge is crucial for designing physical activity programs tailored and adapted to the level of metabolic impairment and age of obese patients. The hypothesis is that mechanical overload associated with obesity has positive effects on torque production in the absence of metabolic alteration and the effect of aging but negative effects on fatigability, mainly due to muscular factors; the insulin resistance increases peripheral fatigue (due to an alteration in the excitability of the sarcolemma during fatiguing exercise), central fatigue, and slows recovery; the development of inflammation and lipid infiltration, which are more pronounced in obese subjects, further affect torque production through inhibition of the nervous control and alteration of contractile properties and muscle architecture, all these phenomena leading to a decrease in torque production and increased fatigability, cumulating with the effects of the ageing (sarcopenia).

DETAILED DESCRIPTION:
The limited data available in the literature suggest that insulin resistance, low-grade inflammation and muscle lipid infiltration may negatively impact torque production capacity and promote neuromuscular fatigability. Insulin resistance thus has effects on blood perfusion of active muscles, via effects on the autonomic nervous system (Petrofsky and al. 2009). Insulin resistance is also associated with a disruption of Na+/K+ pump activity, excitation-contraction coupling, intracellular ATP concentration (Orlando and al. 2016) and mitochondrial function (Slattery and al. 2014). All these effects are expected to increase the development of peripheral fatigue in obese patients with type 2 diabetes and impaired mitochondrial function is expected to result in impaired post-exercise recovery capacity. Inflammation can also affect the torque production. Some studies have shown a negative correlation between muscle torque production and inflammatory status in obese adolescents (Ruiz and al. 2008) and seniors (Visser and al. 2002). Inflammation is associated with reduced muscle mass, which may result from inhibition of protein synthesis (Guillet and al. 2012). Inflammation could also have negative effects on the nervous factors of torque production, via the stimulation of afferences III and IV, as suggested in the healthy subject (Dousset and al. 2007). However, this has never been demonstrated. Finally, oedema associated with the inflammatory reaction could modify the architecture and muscle dimensions, as demonstrated in healthy subjects (Ishikawa and al. 2006) or those suffering from inflammatory diseases (Kaya and al. 2013). To date, the consequences of low-grade inflammation, combined or not with aging, on the muscle and nervous factors of force production in obese adults have yet to be characterized experimentally. Muscle lipid infiltration can also have negative effects on muscle protein synthesis (Tardif and al. 2014) and especially on strength. This has been frequently reported in non-obese elderly people (Sipilä and Suominen 1994). Interestingly, another study reported a negative correlation between intramuscular lipid content and level of quadriceps voluntary activation in non-obese elderly people (Yoshida and al. 2012), which may explain the correlation discussed above. To our knowledge, no data are available for adult obese patients. However, it can be assumed that lipid infiltration would have inhibitory effects on the level of activation of motor units, and therefore on the production of force. It is also likely that lipid infiltration limits muscle architectural adaptations to overweight (contractile and adipose tissues competing to develop in a restricted muscle volume). Mathematical modelling of the effects of lipid infiltration on muscle mechanics (Rahemi and al. 2015) suggests that intramuscular lipids could disrupt contractile activity by limiting the shortening of muscle fascicles, and transverse muscle deformation during muscle contraction. However, these theoretical predictions have yet to be confirmed by experimental data.

The PLANEUROB research project is a physiological observational study comparing the respective effects of mechanical overload, metabolic disorders and age on torque production, fatigability and functional capacity in obese people. Subjects will have to perform a fatigue protocol, an adapted Margaria test and a 6 minutes walking test in one session. Blood samples, muscular ultrasound scanner and physical activity assessment will also be achieved.

Data will be analysed using LabChart 7.3 Pro software (ADInstrument, New South Wales, Australia), ImageJ (NIH Image, Bethesda, Maryland, USA) and Statistica 8.0 software (StatSoft, Inc.) and significance will be accepted at a two-sided alpha level of p<.05. The normality and homogeneity of the variables will be checked respectively from a Shapiro- Wilk test and a Barlett test. If normality and homogeneity of the variables are verified, absolute values of variables (Torque, EMG, mean grey, etc.) will be compared using two factors (age x metabolic disorders) analyses of variance (ANOVA) with repeated measures. If analyses reveal a significant effect of any factor or interaction of factors, post-hoc Newman-Keuls tests will be performed to determine differences between the different conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject, aged between 20 and 70 years old (inclusive terminals).
* Subject with a BMI greater than 30kg/m².
* Subject with a stable weight for at least 3 months before the start of the study.
* Subject capable and willing to comply with the protocol and willing to give informed consent in writing.
* Subject affiliated to a social security system.

Exclusion Criteria:

Subject with a medical or surgical history deemed by the investigator to be incompatible with the study.

* Subject with a medical contraindication to intense activity.
* Subject weighing more than 170kg, which may damage the dynamometer chair.
* Subject with a treatment that, in the investigator's opinion, may interfere with the evaluation of study criteria, period of exclusion from a previous clinical study.
* Subject who has received a total amount of compensation since the beginning of the calendar year, greater than 4500 euros (amount may change depending on the regulation).
* Subject with a linguistic or physiological disability to sign informed consent.
* Subject deprived of liberty by administrative of juridical decision, under guardianship or curatorship.
* Pregnant or breastfeeding women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Maximal torqueof the knee extensors (in N.m) | day 7
  Maximal torque of the knee extensors (in N.m) measured with a dynamometer.
Fatiguability of the knee extensors (in N.m) | day 7
  Fatiguability of the knee extensors (in N.m) measured with a dynamometer.

SECONDARY OUTCOMES:
Maximal muscle power of the lower limb | day 1
  Maximal muscle power of the lower limb muscles measured during an adapted Margaria test (15 steps by walking).
Functional capacity | day 1
  Functional capacity assessed by a 6 minutes walking test.
Muscle contractile properties | day 7
  Muscle contractile properties using muscle twitches and the doublet torque amplitude (100Hz, in N.m) measured using electrical muscle stimulation.
Measure of alteration of the excitation contraction coupling | day 7
  Alteration of the excitation contraction coupling using the high frequency (100Hz)/ low frequency (10Hz) ratio evoked by electrical muscle stimulation.
Measure of Sarcolemma excitability | day 7
  Sarcolemma excitability using muscle action potential amplitude (i.e M-wave, in mV) evoked by electrical muscle stimulation and measured by surface electromyography (EMG).
Measure of Voluntary activation level (%) | day 7
  Voluntary activation level (%) assessed by using the twitch interpolation technique.
Measure of Fascicule length (mm), | day 1
  Fascicule length (mm) measured by B-mode real time ultrasound scanner.
Measure of pennation angle (degree) | day 1
  pennation angle (degree) measured by B-mode real time ultrasound scanner.
Measure cross-sectional area (cm²) | day 1
  cross-sectional area (cm²) measured by B-mode real time ultrasound scanner.
Measure muscular lipid infiltration (%) | day 1
  muscular lipid infiltration (%) measured by B-mode real time ultrasound scanner.
Measure of Glycemia (g/L) | day 1
  Glycemia in blood samples.
Measure of insulinemia (pmol/L) | day 1
  insulinemia in blood samples.
Measure of HbA1c(mmol/mol) | day 1
  HbA1c in blood samples.
Measure of triglyceridemia (g/L) | day 1
  triglyceridemia in blood samples.
Measure of CRP (mg/L) | day 1
  CRP in blood samples.
Height in cm | day 1
  Anthropometric measure of height
weight in kg | day 1
  Anthropometric measure of weight
waist circumference in cm | day 1
  Anthropometric measure of waist circumference.
Physical activity | day 1
  Physical activity measured with Global Physical Activity Questionnaire
Physical activity | day 1
  Physical activity measured with Physical Activity Questionnaire
Physical activity | day2, day 3, day 4, day 5, day 6
  Physical activity measured accelerometery.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France